CLINICAL TRIAL: NCT04455503
Title: A Phase 1/2, Study of Adjuvant Immunotherapy With EVX-02 and Anti-PD-1 After Complete Resection of Stage IIIB/IIIC/IIID or Stage IV Melanoma in Patients at High Risk for Recurrence
Brief Title: Study of Adjuvant Immunotherapy With EVX-02 and Anti-PD-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on the promising interim results of study part 1, it was decided to further accelerate the development of the 2nd generation DNA plasmid immunotherapy. Therefore enrolment of patients was completed after study part 1
Sponsor: Evaxion Biotech A/S (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVX-02-001
Record Dates: First submitted 2020-06-14; First posted 2020-07-02 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Melanoma Stage IV; Melanoma Stage III
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: Nivolumab and EVX-02A (Experimental): EVX-02A administered IM.
  Interventions: Drug: EVX-02A
- Cohort B: Nivolumab and EVX-02B (Experimental): EVX-02B administered IM.
  Interventions: Drug: EVX-02B
- Cohort C: Nivolumab and EVX-02A OR Nivolumab and EVX-02B (Experimental): The selected delivery methodology either EVX02A or EVX-02B.
  Interventions: Drug: EVX-02A OR EVX-02B

INTERVENTIONS:
Drug: EVX-02A — Up to 8 patients will receive EVX-02A administered IM.
  Other Names: A
  Arms: Cohort A: Nivolumab and EVX-02A
Drug: EVX-02B — Up to 8 patients will receive EVX-02B administered IM.
  Other Names: B
  Arms: Cohort B: Nivolumab and EVX-02B
Drug: EVX-02A OR EVX-02B — EVX-02A or EVX-02B will be used. Patients: 24 to 30
  Other Names: C
  Arms: Cohort C: Nivolumab and EVX-02A OR Nivolumab and EVX-02B

SUMMARY:
This is a Phase 1/2, open label, multi-centre study to assess the safety, tolerability, PD, and efficacy of adjuvant immunotherapy EVX-02 vaccine and anti-PD-1 (Nivolumab) in patients who have had a complete resection of a Stage IIIB/IIIC/IIID or Stage IV melanoma who are at high risk of recurrence.

DETAILED DESCRIPTION:
This study will be conducted in two parts: a safety, efficacy and PD response part using two different drug delivery methods and an expansion cohort.

All patients will be administered with anti-PD-1 once every 4 weeks for up to 1 year commencing on Day 1 and with EVX-02 vaccine as soon as it is produced.

Part 1 will consist of two cohorts:

Cohort A: Will receive EVX- 02A delivered by delivery methodology 1. Cohort B: Will receive EVX- 02B delivered by delivery device 2. Part 2 (Cohort C) will be an expansion cohort. In this part, only one delivery methods, either EVX-02A or EVX-02B with will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written ICF prior to performing any protocol-related procedures, which are not part of normal standard care.
2. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, tumour sample including core needle biopsy as required, and other requirements of the study.
3. Male or female ≥ 18 years of age at the time of informed consent.
4. Stage IIIB/IIIC/IIID or Stage IV AJCC (8th edition) (AJCC, 2018) before complete resection.

   Please note: If Stage III melanoma (whether Stage IIIB or IIIC or IIID) the patients must have clinically detectable lymph nodes that are confirmed as malignant on the pathology report and/or ulcerated primary lesions, and/or in transit metastasis. The pathology report must be reviewed, signed and dated by the Investigator; this process must be done prior to enrolling patients into the study. Clinically detectable lymph nodes are defined as:
   1. a palpable node (confirmed as malignant by pathology) after the CLND
   2. a non-palpable but enlarged lymph node by CT scan (at least 15 mm in short axis) and confirmed as malignant by pathology after the CLND
   3. a PET scan positive lymph node of any size confirmed by pathology after CLND
   4. evidence of pathologically macro metastatic disease in one or more lymph nodes defined by one or more foci of melanoma at least 1 cm in diameter If Stage IV melanoma, the pathology report confirming negative margins must be reviewed, dated, and signed by the Investigator prior to randomisation.
5. Cutaneous Melanoma, with metastases to regional lymph nodes or distant metastases, or in transit metastases, that can be surgically resected with negative margin on resected specimens.
6. Specimen from the resected tumour tissue must be provided for evaluation by NGS.
7. ECOG performance status score of 0 or 1.
8. Screening laboratory values must meet the following criteria and must be reconfirmed for eligibility within 72 hours prior to first dose of anti-PD-1 on Day 1:

   i. WBCs ≥ 2000/μL (2.0 x 109/L) ii. Neutrophils ≥ 1500/μL (1.5 x109/L) iii. Platelets ≥ 100 x 10³/μL (100 x 109/L) iv. Haemoglobin ≥ 9.0 g/dL (90 g/L) v. Creatinine Serum creatinine ≤ 1.5 x ULN or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula) vi. AST ≤ 3 x ULN vii. ALT ≤ 3 x ULN viii. Total Bilirubin ≥ 1.5 x ULN (except patients with Gilbert Syndrome who must have total bilirubin < 3.0 mg/dL)
9. Life expectancy > 6 months at Screening.
10. WOCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
11. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of hCG]) within 24 hours prior to first dose of anti-PD-1 on Day 1.
12. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug plus 30 days (duration of ovulatory cycle). The half-life of nivolumab is up to 25 days. WOCBP should therefore use an adequate method to avoid pregnancy for a total of 23 weeks post-treatment completion.
13. Men who are sexually active with a WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of the study drug(s) plus 90 days (duration of sperm turnover). The half-life of nivolumab is up to 25 days, men should therefore use an adequate method of contraception for a total of 31 weeks post-treatment completion.
14. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However, WOCBP must still undergo pregnancy testing.
15. Disease-free at study enrolment (after surgery) based upon pathology report review by the Investigator.

Exclusion Criteria:

1. Known or active other malignancies that have needed treatment (excluding palliative radiation) within 2 years prior to Cycle 1 Day 1 are excluded except for the following:

   1. Curatively resected non-melanomatous skin cancer
   2. Curatively treated cervical carcinoma in situ
   3. Non-metastatic breast and prostate cancer patients with stable disease > 12 months
   4. Other stable malignancies may be permitted based on case-by-case discussions with Sponsor and Medical Monitor approval.
2. Patients with clinically occult lymph nodes (i.e. detected by SLN biopsy) stage N1a and N2a.
3. Participated in any other investigational study, unless treatment in that study has been discontinued at least 30 days or period of five half-lives prior to Screening.
4. Known or suspected allergy or hypersensitivity to any of the therapeutic agents to be administered during the study.
5. Uncontrolled concurrent illness including, but not limited to, active infection, symptomatic congestive heart failure or cardiac arrhythmia.
6. Has a history of clinically significant GI disease, renal, hepatic, neurologic, haematologic, endocrine, oncologic, pulmonary, immunologic, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardise the safety of the patient or impact the validity of the study results.
7. Uncontrolled mental disease or psychotic manifestation that, in the opinion of the Investigator, would prohibit compliance with the protocol, the understanding of the ICF, or the ability to withdraw from the study.
8. Known history of or positive test for HIV or known immunodeficiency syndrome (AIDS).
9. For patients with evidence of chronic HBV infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
10. Patients with a history of HCV infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
11. Pregnant or nursing women.
12. Ocular or uveal melanoma.
13. History of carcinomatosis meningitis.
14. History of Grade ≥ 3 allergy to human monoclonal antibodies.
15. Active, known, or suspected autoimmune disease or immunosuppressive conditions with the exception of vitiligo, type 1 diabetes, residual autoimmune-related hypothyroidism requiring hormone replacement, or psoriasis not requiring systemic treatment.
16. Prior treatment with immune-modulatory agents including, but not limited to: IL-2, CTLA-4 blockade, PD-1/PD-L1 blockade, CD40 stimulation, CD137 stimulation - with the exception of IFN-α given as adjuvant treatment for high risk, surgically resected melanoma (Note. IFN-α therapy must have been discontinued more than 4 weeks prior to enrolment in the study).
17. Prior investigational melanoma-directed cancer vaccine therapy.
18. Prior chemotherapy, including targeted therapy such as BRAF or MEK inhibition.
19. Use of a non-oncology vaccine therapy for prevention of infectious diseases up to 4 weeks prior to enrolment in the study.
20. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to first dose of anti-PD-1 on Day 1. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) | Measurements at Baseline through study completion, an average of 1 year
  Measure through CTCAE version 5.0
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- blood pressure | Measurements at Baseline through study completion, an average of 1 year
  Measured by result of the Vital Sign- blood pressure
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign-heart rate | Measurements at Baseline through study completion, an average of 1 year
  Measured by result of the Vital Sign- heart rate
Safety and tolerability (Incidence of Treatment-Emergent Adverse Events) measure through Physical exam | Measurements at Baseline through study completion, an average of 1 year
  Measured by result of the physical exam which includes general appearance, skin, eyes/ears/nose/throat, head and neck.
Pharmacodynamic response (PD) of EVX-02 assessed by IFN-y ELISPOT | Measurements at Baseline through study completion, an average of 1 year
  The pharmacodynamic (PD) response of EVX-02 will be assessed by detecting vaccine induced circulating neoepitope-specific T cells. Blood samples will be collected prior, during and after immunization and the immunotherapy induced T cell responses will be assayed by IFN-y ELISPOT.
Pharmacodynamic response (PD) of EVX-02 assessed by MHC I multimer analysis | Measurements at Baseline through study completion, an average of 1 year
  The pharmacodynamic (PD) response of EVX-02 will be assessed by detecting vaccine induced circulating neoepitope-specific T cells. Blood samples will be collected prior, during and after immunization. The samples will be analyzed by MHC I multimer analyses detecting neoepitope-recognizing CD8+ T cells reported as frequencies of positive cell out of CD8+ T cells.
Pharmacodynamic response (PD) of EVX-02 by intracellular cytokine staining and flow cytometry | Measurements at Baseline through study completion, an average of 1 year
  The pharmacodynamic (PD) response of EVX-02 will be assessed by detecting vaccine induced circulating neoepitpe-specific T cells. Blood samples will be collected prior, during and after immunization. The samples will be analysed by flow cytometry to detect vaccine induced intracellular cytokine response, reported as frequencies of neoepitope-reactive CD4+ cells and CD8+ T cells.

SECONDARY OUTCOMES:
Efficacy measure through Relapse-free survival (RFS) | Measurements at Baseline through study completion, an average of 1 year
  Measured by result of Relapse-free survival (RFS)

OTHER OUTCOMES:
PD response of EVX-02 assessed by monitoring the quantity of cfDNA in plasma | Measured at Screening, Day -84 to Day -1, Day 1, Day 84, Day 168, Day 252, Day 336 and early termination
  To monitor the plasma level cfDNA, blood sample will be obtained prior, during and after treatment with EVX-02 and the fluctuations of the level cfDNA will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bavanthi Balakrishnar, Principal Investigator — Liverpool Hospital
Locations (6):
- Australia (6):
  - Liverpool Hospital, Goulburn, New South Wales
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Ballarat Health Services, Drummond, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Cancer Trials, Nedlands, Western Australia